CLINICAL TRIAL: NCT05005702
Title: Effects of Inspiratory Muscle Training on Functional Capacity in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0301 Ayesha Fatima
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Patients were assigned to inspiratory muscle training (IMT) for 6 weeks. During training, patients were instructed to maintain diaphragmatic breathing, and try to maintain 10-15 breaths, and rested 5-10 between breaths. As soon as the patients managed; they were encouraged to maintain 25-30 breaths at each workload. All patients wore nose-clip during training. The inspiratory load was set at 40% of maximal inspiratory pressure. The training session was supervised at the hospital.
  Interventions: Other: Inspiratory Muscle training

INTERVENTIONS:
Other: Inspiratory Muscle training — Patients received IMT for 30-minute per day, 3 days per week for 3 weeks using the Threshold Inspiratory Muscle training device (product Phillips). During training, patients were instructed to maintain diaphragmatic breathing, and try to maintain 10-15 breaths, and rested 5-10 between breaths. As soon as the patients managed; they were encouraged to maintain 25-30 breaths at each workload. All patients wore nose-clip during training.
  Inspiratory muscle training diaries were checked weekly. The inspiratory load was set at 40%of maximal inspiratory pressure.

SUMMARY:
Heart failure is a complex clinical syndrome manifesting as inability to supply adequate blood flow throughout the body due to any structural or functional cardiac abnormality. The most common complaints are exercise intolerance, balance, dyspnea, and fatigue in patients with heart failure. It is clearly stated that pulmonary muscle weakness is prevalent and contributes to exercise intolerance in patients with heart failure. Purpose of the study was to evaluate the efficacy of inspiratory muscle traning on pulmonary muscle strength, pulmonary function test, functional capacity and quality of life. The tools used were 6-minute walk test, spirometry, IMT threshold device for IMT strength, and Quality of life. Study was conducted in 20 patients in single group and pre and post values were evaluated. The significance this study bears was that it helped defining for us that to how much extent we can improve the physical and pulmonary functional capacity using inspiratory muscle training. Data were analysed using spss 22.0.mean and standard deviation were calculated. Appropirate the stasitical test were used after checking normailty of data. Parametric test were used for data analysis using SPSS 22

ELIGIBILITY:
Inclusion Criteria:

1. Adults 40-60 years old who are sedentary.
2. Left ventricular ejection fraction of less than 45% evaluated by echocardiogram
3. Functional class II and III (New York Heart Association)
4. FEV1 less than 80%, predicted and/or FEV1/ forced vital capacity (FVC) ratio of more than 70% predicted, and clinical stability.
5. Ex-smokers of more than 5 years.

Exclusion Criteria:

1. Myocardial infarction
2. Complex arrhythmias
3. Uncontrolled hypertension
4. Angina pectoris.
5. Cognitive disorders
6. Recent any trauma.
7. Chronic respiratory disease.
8. Unstable angina
9. Recent viral infections (6 months before the study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test (6MWT) Distance | 6 week
  Six-minute walk test (6MWT) was applied in a 30-m unobstructed corridor. Patients and controls were instructed to walk at their own pace but to cover as much meter as possible within 6 min. Each minute standardized encouragement was given to the patients. Patients were allowed to stop and rest during the test but were instructed to go on walking as soon as they were able to do so. Heart rate and spo2 were monitored using pulse oximetry before and ending the test. Maximum heart rate values achieved during the tests were recorded. The rate of the perceived exertional scale was used before and after the 6MWT. The 6MWT distance is expressed as a percentage of the predicted values.
Pulmonary function test. | 6 week
  Measurements of forced vital capacity and forced expiratory volume in 1, forced expiratory volume in one second/forced vital capacity, peak expiratory pressure was obtained with a computerized spiro-lab device as recommended by the European respiratory society, and results were expressed as a percentage of predicted values.
SF-36 | 6 week
  Quality of life was assessed using SF-36. The SF-36 is a generic measure, consisting of eight
  subscales and 36 items. These subscales are physical functioning, role-physical, role- emotional, mental health, social functioning, bodily pain, general health. All subscales range
  from 0 (worst possible) to100 points (best health).

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zayed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savci S, Degirmenci B, Saglam M, Arikan H, Inal-Ince D, Turan HN, Demircin M. Short-term effects of inspiratory muscle training in coronary artery bypass graft surgery: a randomized controlled trial. Scand Cardiovasc J. 2011 Oct;45(5):286-93. doi: 10.3109/14017431.2011.595820. Epub 2011 Jul 27. PMID 21793631
- [Background] Leite JC, Brandao DC, Brandao SCS, Fuzari HKB, Vidal TM, Frutuoso J, Remigio MI, de Araujo BTS, Campos SL, Dornelas de Andrade A. Effectiveness of inspiratory muscle training associated with a cardiac rehabilitation program on sympathetic activity and functional capacity in patients with heart failure: a study protocol for a randomized controlled trial. Trials. 2020 Jun 12;21(1):519. doi: 10.1186/s13063-020-04363-6. PMID 32532283
- [Background] Marco E, Ramirez-Sarmiento AL, Coloma A, Sartor M, Comin-Colet J, Vila J, Enjuanes C, Bruguera J, Escalada F, Gea J, Orozco-Levi M. High-intensity vs. sham inspiratory muscle training in patients with chronic heart failure: a prospective randomized trial. Eur J Heart Fail. 2013 Aug;15(8):892-901. doi: 10.1093/eurjhf/hft035. Epub 2013 Mar 19. PMID 23512093
- [Background] Dall'Ago P, Chiappa GR, Guths H, Stein R, Ribeiro JP. Inspiratory muscle training in patients with heart failure and inspiratory muscle weakness: a randomized trial. J Am Coll Cardiol. 2006 Feb 21;47(4):757-63. doi: 10.1016/j.jacc.2005.09.052. Epub 2006 Jan 26. PMID 16487841
- [Background] Cordeiro ALL, Mascarenhas HC, Landerson L, Araujo JDS, Borges DL, Melo TA, Guimaraes A, Petto J. Inspiratory Muscle Training Based on Anaerobic Threshold on the Functional Capacity of Patients After Coronary Artery Bypass Grafting: Clinical Trial. Braz J Cardiovasc Surg. 2020 Dec 1;35(6):942-949. doi: 10.21470/1678-9741-2019-0448. PMID 33113311
- [Background] Arena R, Cahalin LP, Borghi-Silva A, Phillips SA. Improving functional capacity in heart failure: the need for a multifaceted approach. Curr Opin Cardiol. 2014 Sep;29(5):467-74. doi: 10.1097/HCO.0000000000000092. PMID 25036108
- [Background] Winkelmann ER, Chiappa GR, Lima CO, Viecili PR, Stein R, Ribeiro JP. Addition of inspiratory muscle training to aerobic training improves cardiorespiratory responses to exercise in patients with heart failure and inspiratory muscle weakness. Am Heart J. 2009 Nov;158(5):768.e1-7. doi: 10.1016/j.ahj.2009.09.005. Epub 2009 Oct 2. PMID 19853695
- [Background] Fernandez-Rubio H, Becerro-de-Bengoa-Vallejo R, Rodriguez-Sanz D, Calvo-Lobo C, Vicente-Campos D, Chicharro JL. Inspiratory Muscle Training in Patients with Heart Failure. J Clin Med. 2020 Jun 2;9(6):1710. doi: 10.3390/jcm9061710. PMID 32498445
- [Background] de Abreu RM, Rehder-Santos P, Minatel V, Dos Santos GL, Catai AM. Effects of inspiratory muscle training on cardiovascular autonomic control: A systematic review. Auton Neurosci. 2017 Dec;208:29-35. doi: 10.1016/j.autneu.2017.09.002. Epub 2017 Sep 7. PMID 28916152
- [Background] Zeren M, Demir R, Yigit Z, Gurses HN. Effects of inspiratory muscle training on pulmonary function, respiratory muscle strength and functional capacity in patients with atrial fibrillation: a randomized controlled trial. Clin Rehabil. 2016 Dec;30(12):1165-1174. doi: 10.1177/0269215515628038. Epub 2016 Jan 27. PMID 26817809
- [Background] Hermes BM, Cardoso DM, Gomes TJ, Santos TD, Vicente MS, Pereira SN, Barbosa VA, Albuquerque IM. Short-term inspiratory muscle training potentiates the benefits of aerobic and resistance training in patients undergoing CABG in phase II cardiac rehabilitation program. Rev Bras Cir Cardiovasc. 2015 Jul-Aug;30(4):474-81. doi: 10.5935/1678-9741.20150043. PMID 27163422
- [Background] Sadek Z, Salami A, Joumaa WH, Awada C, Ahmaidi S, Ramadan W. Best mode of inspiratory muscle training in heart failure patients: a systematic review and meta-analysis. Eur J Prev Cardiol. 2018 Nov;25(16):1691-1701. doi: 10.1177/2047487318792315. Epub 2018 Aug 3. PMID 30073849
- [Background] Ramalho SHR, Cipriano Junior G, Vieira PJC, Nakano EY, Winkelmann ER, Callegaro CC, Chiappa GR. Inspiratory muscle strength and six-minute walking distance in heart failure: Prognostic utility in a 10 years follow up cohort study. PLoS One. 2019 Aug 1;14(8):e0220638. doi: 10.1371/journal.pone.0220638. eCollection 2019. PMID 31369636